CLINICAL TRIAL: NCT02291458
Title: The Effect of L-arginine on Brown Adipose Tissue Metabolism in South Asian and White Caucasian Subjects
Brief Title: L-arginine and Brown Adipose Tissue
Acronym: ArgMB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NL2014-001733-86
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Adipose Tissue, Brown; Glucose Intolerance; Nitric Oxide
MeSH Terms: conditions — Glucose Intolerance | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-arginine (Experimental): Subjects will receive 9 gram of L-arginine per day in three gifts (3dd 3 gram) during 6 weeks.
  Interventions: Drug: L-arginine
- Placebo (Placebo Comparator): Subjects will receive 9 gram of placebo per day in three gifts (3 dd 3 gram) during 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-arginine — 9 gram L-arginine / day for 6 weeks
  Other Names: Argimax
  Arms: L-arginine
Drug: Placebo — 9 gram placebo / day for 6 weeks
  Arms: Placebo

SUMMARY:
The South Asian population is facing an epidemic of type 2 diabetes, of which the underlying cause is still unknown. It is currently hypothesized that an ethnic susceptibility towards a disturbed energy metabolism may underlie this disadvantageous metabolic phenotype. In line with this, the investigators recently discovered that Dutch South Asian subjects have 32% lower resting energy expenditure (REE) and 34% lower energy-combusting brown adipose tissue (BAT) compared to matched white Caucasians. Nitric oxide (NO) was recently shown to be crucial for BAT development and, interestingly, South Asians have diminished NO bioavailability. Thus, the disadvantageous metabolic phenotype in South Asians may be caused by diminished NO bioavailability resulting in lower BAT volume. Therefore, the investigators hypothesize that increasing NO generation in the body by administration of L-arginine, the precursor of NO, will improve their metabolic phenotype by increasing BAT volume, thereby increasing REE and clearance of triglycerides and glucose by BAT. To investigate this, the investigators will perform a randomized placebo-controlled multicenter cross-over study in moderately obese Dutch South Asians and matched white Caucasians. Subjects will receive L-arginine (9 gram/day) or placebo for 6 weeks, followed by a wash-out period of 4 weeks and then again 6 weeks of one of either treatments. At the end of both treatment periods, a cold-induced PET-CT scan will be performed. Furthermore, muscle and fat biopsies will be obtained and thermoregulation will be assessed.

DETAILED DESCRIPTION:
Rationale: The South Asian population originally descends from the Indian subcontinent and represents approximately 20% of the total world population. This population is facing an epidemic of type 2 diabetes, of which the underlying cause is still unknown. A high prevalence of a disadvantageous metabolic phenotype, consisting of obesity, insulin resistance and dyslipidemia, may at least in part contribute to this excess risk. It is currently hypothesized that an ethnic susceptibility towards a disturbed energy metabolism may underlie this disadvantageous metabolic phenotype. In line with this, the investigators recently discovered that Dutch South Asian subjects have 32% lower resting energy expenditure (REE) and 34% lower energy-combusting brown adipose tissue (BAT) compared to matched white Caucasians. Nitric oxide (NO) was recently shown to be crucial for BAT development and, interestingly, South Asians have diminished NO bioavailability. Thus, the disadvantageous metabolic phenotype in South Asians may be caused by diminished NO bioavailability resulting in lower BAT volume. Therefore, the investigators hypothesize that increasing NO generation in the body by administration of L-arginine, the precursor of NO, will improve their metabolic phenotype by increasing BAT volume, thereby increasing REE and clearance of triglycerides and glucose by BAT.

Objectives: The primary objectives are: 1) to determine the effect of L-arginine on glucose uptake by brown adipose tissue and to assess whether the effect differs between South Asian and white Caucasian subjects; 2) to determine the effect of L-arginine on whole body energy expenditure and to assess whether the effect differs between South Asian and white Caucasian subjects; 3) to determine the effect of L-arginine on fat mass and to assess whether the effect differs between South Asian and white Caucasian subjects.

Study design: A randomized placebo-controlled multicenter cross-over study will be performed in moderately obese Dutch South Asians and matched white Caucasians. Subjects will receive L-arginine (9 gram/day) or placebo for 6 weeks, followed by a wash-out period of 4 weeks and then again 6 weeks of one of either treatments. At the end of both treatment periods, a cold-induced PET-CT scan will be performed. Furthermore, muscle and fat biopsies will be obtained, thermoregulation will be assessed, an oral glucose tolerance will be performed and the investigators will assess NO-dependent and independent vasodilation by means of iontophoresis.

Study population: Mildly obese (BMI 25-30 kg/m2) pre-diabetic male volunteers of South Asian and white Caucasian descent aged between 35-50 years.

Intervention: The intervention will consist of administration of 9 grams of L-arginine per day in three gifts (3dd 3 gram).

ELIGIBILITY:
Inclusion Criteria:

* Caucasian or South Asian ethnicity
* Age: 35-50 years
* Gender: male
* BMI: 25-30 kg/m2
* Plasma glucose levels 2 h after OGTT between 7.8 and 11 mM (e.g. impaired glucose tolerance) or Fasting plasma glucose levels > 5.5 mM
* Good general health

Exclusion Criteria:

* Type 2 diabetes (determined on basis of oral glucose tolerance test (OGTT))
* BMI > 30 kg/m2
* Plasma glucose levels 2 h after OGTT < 7.8 mM
* Plasma L-arginine levels < 41 or > 114 uM
* Use of beta-blockers (these inhibit BAT activity) < 1 month before start of study or during study
* Systolic blood pressure < 90 mmHg
* Haematocrit < 0.41 or > 0.51 l/l
* Haemoglobin < 8.5 or > 11.0
* Creatinine (enzymatic method) < 45 or > 100 μmol/L
* ASAT > 45 U/L
* ALAT > 50 U/L
* Alkaline phosphatase > 125 U/L
* Gamma GT > 45 U/L
* Participation in an intensive weight-loss program or vigorous exercise program during the last year before the start of the study
* Abuse of drugs and/or alcohol
* Hyperthyroidism or hypothyroidism
* Participation in earlier research or medical examinations that included PET-CT scanning
* Psychologically unstable subjects (as judged by the treating medical specialist)
* Subjects with mental retardation (as judged by the treating medical specialist)
* Subjects with severe behaviour disorders (as judged by the treating medical specialist)

Ages: 35 Months to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Standard uptake value of Brown adipose tissue | 6 weeks
  Glucose uptake by brown adiopse tissue will be assessed by cold-induced 18F-FDG PET-CT scan
Energy expenditure | 6 weeks
  Energy expenditure will be determined by means of indirect calorimetrie
Fat mass | 6 weeks
  Fat mass will be determined by DEXA scan

SECONDARY OUTCOMES:
Body temperatures | 6 weeks
  Skin and core body temperatures as well as gradients will be assessed by means of iButtons and ingestion of a telemetric pill, respectively.
Skin perfusion and endothelial-dependent and independent vasodilation | 6 weeks
  This will be measured by means of Laser Doppler Flowmetry (LDF) and iontophoresis
Skeletal muscle mitochondrial respiration/uncoupling | 6 weeks
  This will be determined in muscle biopsies by using the Oroboros 2k Oxygraph instrument present in our laboratory .
Brown adipocyte recruitment and inflammation in WAT | 6 weeks
  This will be measured in subcutaneous WAT biopsies by assessing mRNA expression via real time polymerase-chain reaction (RT-PCR) and protein content by immunohistochemical stainings.
Blood parameters | 6 weeks
  Venous blood will be drawn by means of a catheter placed in the antecubital vein of the underarm. By using radioimmunoassay, high performance liquid chromotogaphy (HPLC) and enzyme-linked immunosorbent assay (ELISA), blood parameters (i.e. lipids, glucose, inflammatory markers and endothelial activation markers) will be analyzed. In addition, we will perform DNA analyses from blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center +, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Janssen LGM, Van Dam AD, Hanssen MJW, Kooijman S, Nahon KJ, Reinders H, Jazet IM, Van Marken Lichtenbelt WD, Rensen PCN, Appelman-Dijkstra NM, Boon MR. Higher Plasma Sclerostin and Lower Wnt Signaling Gene Expression in White Adipose Tissue of Prediabetic South Asian Men Compared with White Caucasian Men. Diabetes Metab J. 2020 Apr;44(2):326-335. doi: 10.4093/dmj.2019.0031. Epub 2019 Oct 31. PMID 31701693
- [Derived] Boon MR, Hanssen MJW, Brans B, Hulsman CJM, Hoeks J, Nahon KJ, Bakker C, van Klinken JB, Havekes B, Schaart G, Jazet IM, Rensen PCN, van Marken Lichtenbelt WD. Effect of L-arginine on energy metabolism, skeletal muscle and brown adipose tissue in South Asian and Europid prediabetic men: a randomised double-blinded crossover study. Diabetologia. 2019 Jan;62(1):112-122. doi: 10.1007/s00125-018-4752-6. Epub 2018 Oct 30. PMID 30377712
- [Derived] Nahon KJ, Kantae V, den Haan R, Hanssen MJW, Harms AC, van der Stelt M, Hankemeier T, Jazet IM, van Marken Lichtenbelt WD, Rensen PCN, Boon MR. Gene Expression of Endocannabinoid System Components in Skeletal Muscle and Adipose Tissue of South Asians and White Caucasians with Overweight. Obesity (Silver Spring). 2018 Aug;26(8):1332-1337. doi: 10.1002/oby.22245. Epub 2018 Aug 1. PMID 30070030